CLINICAL TRIAL: NCT02532998
Title: A Phase I, Randomized, Single-Blind, Crossover Study to Assess the Pharmacodynamics of AZD9977 Following Single-Dose Administration to Healthy Male Subjects
Brief Title: A Study to Assess the Pharmacodynamic Effect of Single Doses of AZD9977 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: D6400C00004; 2015-002224-11 (EudraCT Number)
Record Dates: First submitted 2015-08-24; First posted 2015-08-26 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Pharmacodynamics; Healthy Subjects
Keywords: Pharmacodynamics; AZD9977; Safety; Tolerability; Pharmacokinetics; Eplerenone; Fludrocortisone
MeSH Terms: interventions — Fludrocortisone; Tablets; Eplerenone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (8):
- Treatment Sequence 1 (Experimental): Period 1: fludrocortisone + eplerenone + AZD9977 Period 2: fludrocortisone + eplerenone + AZD9977 Placebo Period 3: fludrocortisone + AZD9977 Placebo Period 4: fludrocortisone + AZD9977 Period 5: fludrocortisone + eplerenone and/or AZD9977 or AZD9977 Placebo treatment Period 6: fludrocortisone + eplerenone and/or AZD9977 or AZD9977 Placebo treatment
  Interventions: Drug: AZD9977 oral suspension; Drug: AZD9977 placebo oral suspension; Drug: Fludrocortisone, tablets; Drug: Eplerenone, tablets
- Treatment Sequence 2 (Experimental): Period 1: fludrocortisone + AZD9977 Placebo Period 2: fludrocortisone + eplerenone + AZD9977 Period 3: fludrocortisone + AZD9977 Period 4: fludrocortisone + eplerenone + AZD9977 Placebo Period 5: fludrocortisone + eplerenone and/or AZD9977 or AZD9977 Placebo treatment Period 6: fludrocortisone + eplerenone and/or AZD9977 or AZD9977 Placebo treatment
  Interventions: Drug: AZD9977 oral suspension; Drug: AZD9977 placebo oral suspension; Drug: Fludrocortisone, tablets; Drug: Eplerenone, tablets
- Treatment Sequence 3 (Experimental): Period 1: fludrocortisone + AZD9977 Period 2: fludrocortisone + AZD9977 Placebo Period 3: fludrocortisone + eplerenone + AZD9977 Placebo Period 4: fludrocortisone + eplerenone + AZD9977 Period 5: fludrocortisone + eplerenone and/or AZD9977 or AZD9977 Placebo treatment Period 6: fludrocortisone + eplerenone and/or AZD9977 or AZD9977 Placebo treatment
  Interventions: Drug: AZD9977 oral suspension; Drug: AZD9977 placebo oral suspension; Drug: Fludrocortisone, tablets; Drug: Eplerenone, tablets
- Treatment Sequence 4 (Experimental): Period 1: fludrocortisone + eplerenone + AZD9977 Placebo Period 2: fludrocortisone + eplerenone + AZD9977 Period 3: fludrocortisone + AZD9977 Period 4: fludrocortisone + AZD9977 Placebo Period 5: fludrocortisone + eplerenone and/or AZD9977 or AZD9977 Placebo treatment Period 6: fludrocortisone + eplerenone and/or AZD9977 or AZD9977 Placebo treatment
  Interventions: Drug: AZD9977 oral suspension; Drug: AZD9977 placebo oral suspension; Drug: Fludrocortisone, tablets; Drug: Eplerenone, tablets
- Treatment Sequence 5 (Experimental): Period 1: fludrocortisone + eplerenone + AZD9977 Period 2: fludrocortisone + eplerenone + AZD9977 Placebo Period 3: fludrocortisone + AZD9977 Placebo Period 4: fludrocortisone + AZD9977 Period 5: fludrocortisone + eplerenone and/or AZD9977 or AZD9977 Placebo treatment Period 6: fludrocortisone + eplerenone and/or AZD9977 or AZD9977 Placebo treatment
  Interventions: Drug: AZD9977 oral suspension; Drug: AZD9977 placebo oral suspension; Drug: Fludrocortisone, tablets; Drug: Eplerenone, tablets
- Treatment Sequence 6 (Experimental): Period 1: fludrocortisone + AZD9977 Placebo Period 2: fludrocortisone + eplerenone + AZD9977 Period 3: fludrocortisone + AZD9977 Period 4: fludrocortisone + eplerenone + AZD9977 Placebo Period 5: fludrocortisone + eplerenone and/or AZD9977 or AZD9977 Placebo treatment Period 6: fludrocortisone + eplerenone and/or AZD9977 or AZD9977 Placebo treatment
  Interventions: Drug: AZD9977 oral suspension; Drug: AZD9977 placebo oral suspension; Drug: Fludrocortisone, tablets; Drug: Eplerenone, tablets
- Treatment Sequence 7 (Experimental): Period 1: fludrocortisone + AZD9977 Period 2: fludrocortisone + AZD9977 Placebo Period 3: fludrocortisone + eplerenone + AZD9977 Placebo Period 4: fludrocortisone + eplerenone + AZD9977 Period 5: fludrocortisone + eplerenone and/or AZD9977 or AZD9977 Placebo treatment Period 6: fludrocortisone + eplerenone and/or AZD9977 or AZD9977 Placebo treatment
  Interventions: Drug: AZD9977 oral suspension; Drug: AZD9977 placebo oral suspension; Drug: Fludrocortisone, tablets; Drug: Eplerenone, tablets
- Treatment Sequence 8 (Experimental): Period 1: fludrocortisone + eplerenone + AZD9977 Placebo Period 2: fludrocortisone + AZD9977 Period 3: fludrocortisone + eplerenone + AZD9977 Period 4: fludrocortisone + AZD9977 Placebo Period 5: fludrocortisone + eplerenone and/or AZD9977 or AZD9977 Placebo treatment Period 6: fludrocortisone + eplerenone and/or AZD9977 or AZD9977 Placebo treatment
  Interventions: Drug: AZD9977 oral suspension; Drug: AZD9977 placebo oral suspension; Drug: Fludrocortisone, tablets; Drug: Eplerenone, tablets

INTERVENTIONS:
Drug: AZD9977 oral suspension — AZD9977 oral suspension, single dose
Drug: AZD9977 placebo oral suspension — oral suspension, single dose
Drug: Fludrocortisone, tablets — Loading dose of 0.5 mg and maintenance doses of 0.1 mg every second hour up to a total dose of 1.0 mg per treatment period (may be modified to up to 1.3 mg based on emerging data)
Drug: Eplerenone, tablets — 100 mg (2 x 50 mg tablets) single dose, may be modified based on emerging data (will not exceed 500 mg per treatment period)

SUMMARY:
This is a Phase I, Randomized, Single-Blind, Crossover Study to Assess the Pharmacodynamics of AZD9977 following Single-Dose administration to healthy male subjects

DETAILED DESCRIPTION:
This study will be a phase I study to assess the pharmacodynamics of AZD9977 following single-dose administration to healthy male subjects. It is a single-blind (with regards to AZD9977 and AZD9977 Placebo), randomized, four-treatment, four-period crossover design, with a potential 5th and 6th randomized cross-over treatment period. In this study eplerenone is used as a positive control and fludrocortisone will be used as a challenge agent. In addition the safety, tolerability and pharmacokinetics will be assessed.

ELIGIBILITY:
Inclusion criteria

1. Provision of signed and dated written informed consent prior to any study specific procedures.
2. Healthy male subjects aged 18 to 50 years with suitable veins for cannulation or repeated venipuncture.
3. Male subjects must accept to comply with the restrictions for sexual activity provided to them.
4. Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
5. Optional: Provision of signed and dated written informed consent for genetic research.

   Note: Participation in exploratory biomarker research is mandatory. If a subject declines to participate in the genetic component of the study, there will be no penalty or loss of benefit to the subject. The subject will not be excluded from other aspects of the study described in this protocol.
6. Able to understand, read and speak the English language.

Exclusion criteria

1. History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the potential subject at risk because of participation in the study, or influences the results or the potential subject's ability to participate in the study.
2. History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of first dosing with investigational medicinal product (IMP).
4. Any clinically significant abnormalities in hematology, clinical chemistry or urinalysis results, as judged by the investigator.
5. Abnormal findings in vital signs, after 10 minutes resting in the supine position, defined as any of the following:

   * Systolic blood pressure (SBP) < 90 mmHg or ≥ 140 mmHg
   * Diastolic blood pressure (DBP) < 50 mmHg or ≥ 90 mmHg
   * Pulse < 45 or > 85 beats per minute (bpm)
6. Any clinically significant abnormalities on the 12-lead electrocardiogram (ECG), as judged by the investigator.
7. Any positive result at screening for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody, and human immunodeficiency virus (HIV) antibodies.
8. Known or suspected history of drug abuse, as judged by the investigator.
9. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of first dosing. The period of exclusion begins 3 months after the final dose or one month after the last visit whichever is the longest.

   Note: Subjects consented and screened, but not randomized in this study or a previous phase I study, are not excluded.
10. Plasma donation within one month of screening or any blood donation/blood loss > 500 mL during the 3 months prior to screening.
11. History of severe allergy/hypersensitivity or ongoing clinically significant allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD9977.
12. Current smokers or those who have smoked or used nicotine products within the previous 3 months.
13. Positive screen for drugs of abuse, alcohol or cotinine at screening or for each admission to the study center.
14. Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks prior to first dosing.
15. Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during 2 weeks prior to first dosing, or longer if the medication has a long half-life.
16. Known or suspected history of alcohol or drug abuse or excessive intake of alcohol, as judged by the investigator.
17. Involvement of any AstraZeneca or study site employee or their close relatives.
18. Subjects who previously received AZD9977.
19. Judgment by the investigator that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements.
20. Known allergy to eplerenone or fludrocortisone or any of the constituents (including lactose, which is a constituent of Florinef™).
21. History of galactose intolerance.
22. Any infections or at risk of infection (surgery, trauma, or significant infection) within 90 days of screening, or history of skin abscesses within 90 days of screening.
23. Presence, history or family history of long QT syndrome, hypokalemia, hyperkalemia or Torsades de Pointes.
24. Serum potassium < 3.5 mmol/L or ≥ 5.0 mmol/L at screening or for each admission to the study center.
25. Presence or history of active peptic ulcer.
26. History of any psychiatric disorder (including affective, psychotic, behavioral, irritability, anxiety, sleep disturbances and cognitive disorders) which required specialist psychiatric review.
27. Excessive intake of caffeine containing drinks or food (e.g., coffee, tea and chocolate) as judged by the investigator.
28. Subjects who are vegans or have medical dietary restrictions (vegetarians may be included in the study).
29. Subjects who cannot communicate reliably with the investigator.
30. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.
31. In addition, any of the following is regarded as a criterion for exclusion from the genetic research:

    * Previous bone marrow transplant.
    * Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muna Albayaty, MBChB, MSc, MFPM, Principal Investigator — PAREXEL Early Phase Clinical Unit London
Locations (1):
- Research Site, Harrow, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at PAREXEL Early Phase Clinical Unit London, United Kingdom
Pre-assignment Details: This study had a single-blind, randomized, 4-treatment, 4-period crossover design (William's design). A total of 40 participants were enrolled (signed ICF) in this study, of which 23 participants were randomized to receive the study medication.
Groups:
- All Particpants: Twenty three healthy male participants aged 18 to 50 years who satisfied all the study inclusion criteria were included in the study
Period: Overall Study
Arm/Group | All Particpants
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Particpants
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 23

OUTCOME MEASURES:

1. Primary Outcome: Pharmacodynamics of AZD9977 Assessed Per Sodium/Potassium Ratio in Urine in Eplerenone Treatment Versus a Combination Treatment of Eplerenone and AZD9977.
Description: The sum over the urine collection intervals of the logarithm of the urinary sodium/potassium ratio from two hours to eight hours post-dose.
  NOTE: Data are presented as the sum of the difference between ln(Na+) and ln(K+) over the collected intervals 2-4, 4-6 and 6-8 hours.
Time Frame: From 2 hours post dose to 8 hours post dose
Population: The pharmacodynamic (PD) analysis set consisted of all participants in the safety analysis set (SAF) with at least one evaluable sum of the logarithm of the sodium/potassium ratio from two hours up to eight hours post dose, and who had no major protocol deviations thought to impact on the analysis of the PD data.
Measure: Mean (Standard Deviation); unit: sodium/potassium ratio
Groups:
- Treatment C: Participants received fludrocortisone + eplerenone + AZD9977 Placebo.
- Treatment D: Participants received fludrocortisone + eplerenone + AZD9977
Arm/Group | Treatment C | Treatment D
Number analyzed (Participants) | 23 | 23
sodium/potassium ratio | -0.545 (1.19) | 0.694 (1.18)
Statistical Analysis 1: Comparison: Treatment C vs Treatment D; Statistical analysis of urinary sodium/potassium ratio between Treatment C and Treatment D; Test type: Superiority or Other; mixed linear model; Analyses done using mixed linear model involving fixed effect, random effect, and a covariate; Treatment differences = -1.258, 90% CI 2-sided [-1.721 to 0.7945]

2. Secondary Outcome: Observed Maximum Concentration (Cmax) of AZD9977
Description: Pre IMP dose and post IMP dose at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24 hours
Time Frame: From 2 hours post dose to 8 hours post dose
Population: The AZD9977 PK analysis set consisted of all participants who received at least one dose of AZD9977 for whom at least one of the primary PK parameters was evaluable and who had no major protocol deviations thought to impact on the analysis of the AZD9977 PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Groups:
- Treatment B: Participants received fludrocortisone + AZD9977
Arm/Group | Treatment D | Treatment B
Number analyzed (Participants) | 23 | 23
nmol/L | 6238 (16.7) | 5816 (22.2)

3. Secondary Outcome: Area Under Plasma Concentration-time Curve From Zero Extrapolated to Infinity (AUC) of AZD9977.
Description: Pre IMP dose and post IMP dose at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24 hours
Time Frame: From 2 hours post dose to 8 hours post dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | Treatment D | Treatment B
Number analyzed (Participants) | 22 | 21
h*nmol/L | 21060 (18.4) | 19120 (23.9)

4. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to t Hours After Dosing (AUC[0-t]) of AZD9977.
Description: Pre IMP dose and post IMP dose at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24 hours
Time Frame: From 2 hours post dose to 8 hours post dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | Treatment D | Treatment B
Number analyzed (Participants) | 23 | 23
h*nmol/L | 19970 (20.3) | 18520 (23.6)

5. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of AZD9977.
Description: Pre IMP dose and post IMP dose at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24 hours
Time Frame: From 2 hours post dose to 8 hours post dose
Population: The AZD9977 PK analysis set consisted of all subjects who received at least one dose of AZD9977 for whom at least one of the primary PK parameters was evaluable and who had no major protocol deviations thought to impact on the analysis of the AZD9977 PK data.
Measure: Median (Full Range); unit: h
Arm/Group | Treatment D | Treatment B
Number analyzed (Participants) | 23 | 23
h | 0.52 [0.48 to 1.02] | 0.50 [0.48 to 2.50]

6. Secondary Outcome: Terminal Half-life (t½λz) of AZD9977.
Description: Pre IMP dose and post IMP dose at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24 hours
Time Frame: From 2 hours post dose to 8 hours post dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Treatment D | Treatment B
Number analyzed (Participants) | 22 | 21
h | 6.753 (2.322) | 6.726 (1.719)

7. Secondary Outcome: Apparent Clearance (CL/F) of AZD9977.
Description: Pre IMP dose and post IMP dose at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24 hours
Time Frame: From 2 hours post dose to 8 hours post dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Treatment D | Treatment B
Number analyzed (Participants) | 22 | 21
L/h | 23.78 (18.4) | 26.20 (23.9)

8. Secondary Outcome: Apparent Volume of Distribution at Terminal Phase (Vz/F) of AZD9977.
Description: Pre IMP dose and post IMP dose at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24 hours
Time Frame: From 2 hours post dose to 8 hours post dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Treatment B | Treatment D
Number analyzed (Participants) | 21 | 22
L | 246.7 (42.4) | 220.4 (34.3)

9. Secondary Outcome: Apparent Volume of Distribution at Terminal Phase (Vz/F) of Eplerenone.
Description: Pre IMP dose and post IMP dose at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24 hours
Time Frame: From 2 hours post dose to 8 hours post dose
Population: The eplerenone PK analysis set consisted of all participants who received at least one dose of eplerenone for whom at least one of the primary PK parameters was evaluable and who had no major protocol deviations thought to impact on the analysis of the eplerenone PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Treatment C | Treatment D
Number analyzed (Participants) | 23 | 23
L | 49.11 (19.2) | 44.77 (19.3)

10. Secondary Outcome: Apparent Clearance (CL/F) of Eplerenone.
Description: Pre IMP dose and post IMP dose at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24 hours
Time Frame: From 2 hours post dose to 8 hours post dose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Treatment C | Treatment D
Number analyzed (Participants) | 23 | 23
L/h | 10.87 (34.4) | 9.360 (35.9)

11. Secondary Outcome: Terminal Half-life (t½λz) of Eplerenone.
Description: Pre IMP dose and post IMP dose at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24 hours
Time Frame: From 2 hours post dose to 8 hours post dose
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Treatment C | Treatment D
Number analyzed (Participants) | 23 | 23
h | 3.232 (0.8305) | 3.419 (0.8843)

12. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of Eplerenone.
Description: Pre IMP dose and post IMP dose at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24 hours
Time Frame: From 2 hours post dose to 8 hours post dose
Population: as for outcome 9
Measure: Median (Full Range); unit: h
Arm/Group | Treatment C | Treatment D
Number analyzed (Participants) | 23 | 23
h | 1.98 [0.48 to 3.98] | 2.00 [0.97 to 3.98]

13. Secondary Outcome: Observed Maximum Concentration (Cmax) of Eplerenone.
Description: Pre IMP dose and post IMP dose at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24 hours
Time Frame: From 2 hours post dose to 8 hours post dose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment C | Treatment D
Number analyzed (Participants) | 23 | 23
ng/mL | 1557 (26.1) | 1729 (23.2)

14. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to t Hours After Dosing (AUC(0-t)) of Eplerenone.
Description: Pre IMP dose and post IMP dose at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24 hours
Time Frame: From 2 hours post dose to 8 hours post dose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment C | Treatment D
Number analyzed (Participants) | 23 | 23
h*ng/mL | 9035 (33.9) | 10510 (34.6)

15. Secondary Outcome: Area Under Plasma Concentration-time Curve From Zero Extrapolated to Infinity (AUC) of Eplerenone.
Description: Pre IMP dose and post IMP dose at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24 hours
Time Frame: From 2 hours post dose to 8 hours post dose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment C | Treatment D
Number analyzed (Participants) | 23 | 23
h*ng/mL | 9199 (34.4) | 10680 (35.9)

16. Secondary Outcome: Pharmacodynamics of AZD9977 Assessed Per Sodium/Potassium Ratio in Urine in AZD9977 Treatment With Placebo Versus Treatment With AZD9977.
Description: The sum over the urine collection intervals of the logarithm of the urinary sodium/potassium ratio from two hours to eight hours post-dose.
  NOTE: Note: Data are presented as the sum of the difference between ln(Na+) and ln(K+) over the collected intervals 2-4, 4-6 and 6-8 hours.
Time Frame: From 2 hours post dose to 8 hours post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: sodium/potassium ratio
Groups:
- Treatment A: Participants received fludrocortisone + AZD9977 Placebo
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 23 | 23
sodium/potassium ratio | -4.09 (2.11) | -0.694 (1.27)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Statistical analysis of urinary sodium/potassium ratio between Treatment A and Treatment B; Test type: Superiority or Other; mixed linear model; Analyses done using mixed linear model involving fixed effect, random effect, and a covariate; Treatment differences = 3.409, 90% CI 2-sided [2.946 to 3.872]

17. Secondary Outcome: Number of Participants With Clinically Significant Blood Pressure Values.
Description: Clinically significant blood pressure values (if available) were recorded for all participants.
  The systolic blood pressure (mmHg) and diastolic BP (mmHg) was obtained after each subject had rested in the supine position for at least 5 minutes and was performed in accordance with the Schedule of Assessments of study protocol.
  Abnormal findings in blood pressure after 10 minutes resting in the supine position was defined as following:
  * Systolic blood pressure (SBP) < 90 mmHg or ≥ 140 mmHg
  * Diastolic blood pressure (DBP) < 50 mmHg or ≥ 90 mmHg.
Time Frame: From screening to post-study visit, up to 10 weeks
Population: The safety analysis set (SAF) included all participants who received at least one dose of any of the administered products (fludrocortisone, eplerenone or AZD9977/matching placebo) and for whom any safety data post-fludrocortisone dose were available.
Measure: Number; unit: Participants
Arm/Group | Treatment A | Treatment D | Treatment B | Treatment C
Number analyzed (Participants) | 23 | 23 | 23 | 23
Participants | 0 | 0 | 0 | 0

18. Secondary Outcome: Number of Participants With Clinically Significant Pulse Rate.
Description: Clinically significant pulse rate (if available) was recorded for all participants in the study.
  The pulse was obtained after each subject had rested in the supine position for at least 5 minutes and was performed in accordance with the Schedule of Assessments of study protocol.
  Abnormal findings in pulse rate, after 10 minutes resting in the supine position, was defined as following:
  • Pulse < 45 or > 85 beats per minute (bpm)
Time Frame: From screening to post-study visit, up to 10 weeks
Population: The SAF included all subjects who received at least one dose of any of the administered products (fludrocortisone, eplerenone or AZD9977/matching placebo) and for whom any safety data post-fludrocortisone dose were available.
Measure: Number; unit: Participants
Arm/Group | Treatment A | Treatment D | Treatment B | Treatment C
Number analyzed (Participants) | 23 | 23 | 23 | 23
Participants | 0 | 0 | 0 | 0

19. Secondary Outcome: Number of Participants With Clinically Significant Electrocardiogram.
Description: Clinically significant electrocardiogram values were recorded for all participants in the study.
  A 12-lead ECG was obtained after each subject had rested in the supine position for at least 10 minutes and was performed in accordance with the Schedule of Assessments of study protocol.
  The investigator judged the overall interpretation as normal or abnormal. If abnormal, it would have been decided as to whether or not the abnormality was clinically significant and the reason for the abnormality would have been recorded. The investigator could add extra 12-lead resting ECG safety assessments if there were any abnormal findings of if the investigator considered it was necessary for any other safety reason. These assessments would have been entered as an unscheduled assessment.
Time Frame: From screening to post-study visit, up to 10 weeks
Population: The SAF included all participants who received at least one dose of any of the administered products (fludrocortisone, eplerenone or AZD9977/matching placebo) and for whom any safety data post-fludrocortisone dose were available.
Measure: Number; unit: Participants
Arm/Group | Treatment A | Treatment D | Treatment B | Treatment C
Number analyzed (Participants) | 23 | 23 | 23 | 23
Participants | 0 | 0 | 0 | 0

20. Secondary Outcome: Number of Participants With Clinically Significant Physical Examination Values.
Description: Number of participants with clinically significant physical examination values.
  The complete physical examinations included an assessment of the general appearance, respiratory, cardiovascular, abdomen, skin, head, and neck (including ears, eyes, nose, mouth and throat), lymph nodes, thyroid, musculoskeletal and neurological systems. The brief physical examinations included an assessment of the general appearance, skin, abdomen, cardiovascular and respiratory systems. The results of the physical examination were listed by body system for each subject. Body weight was listed by participant and time-point. Any new or aggravated clinically relevant abnormal medical finding at a physical examination as compared with the baseline assessment were reported as an adverse event (AE).
Time Frame: From screening to post-study visit, up to 10 weeks
Population: as for outcome 19
Measure: Number; unit: Participants
Arm/Group | Treatment A | Treatment D | Treatment B | Treatment C
Number analyzed (Participants) | 23 | 23 | 23 | 23
Participants | 0 | 0 | 0 | 0

21. Secondary Outcome: Number of Participants With Clinically Significant Safety Laboratory Tests Values.
Description: Clinically significant safety laboratory test values included hematology, clinical chemistry, urinalysis and urine chemistry, including urine creatinine and uric acid measurements. Viral serology and urine drugs of abuse, alcohol and cotinine were assessed for eligibility. If deterioration in laboratory value was associated with clinical symptoms and/or signs, the symptom or sign were reported as an adverse event and the associated laboratory result was considered as additional information. Laboratory results were listed and summarized according to change from baseline and repeat/unscheduled measurements. Any out of range laboratory results were flagged in the individual listings.
Time Frame: From screening to post-study visit, up to 10 weeks
Population: as for outcome 19
Measure: Number; unit: Participants
Arm/Group | Treatment A | Treatment D | Treatment B | Treatment C
Number analyzed (Participants) | 23 | 23 | 23 | 23
Participants | 0 | 0 | 0 | 0

22. Secondary Outcome: Pharmacodynamics of AZD9977 Assessed by Estimating the Fractional Sodium Excretion in Urine for Each Urine Collection Time Interval.
Description: Pharmacodynamics of AZD9977 by assessment of fractional sodium excretion in urine for each urine collection time interval.
  Pharmacodynamics of AZD9977 after single dosing of AZD9977 with fludrocortisone and/or eplerenone.
Time Frame: From 0 to 8 hours after dosing
Population: The PD analysis set consisted of all participants in the SAF with at least one evaluable sum of the logarithm of the sodium/potassium ratio from two hours up to eight hours post dose, and who had no major protocol deviations thought to impact on the analysis of the PD data.
Measure: Mean (Standard Deviation); unit: % value
Arm/Group | Treatment A | Treatment D | Treatment B | Treatment C
Number analyzed (Participants) | 23 | 23 | 23 | 23
% value
  0 to 2 hours | 0.34 (0.18) | 0.33 (0.19) | 0.32 (0.09) | 0.33 (0.20)
  2 to 4 hours | 0.22 (0.15) | 0.48 (0.21) | 0.35 (0.12) | 0.37 (0.17)
  4 to 6 hours | 0.15 (0.12) | 0.58 (0.19) | 0.36 (0.13) | 0.38 (0.14)
  6 to 8 hours | 0.16 (0.15) | 0.66 (0.23) | 0.36 (0.16) | 0.48 (0.23)

23. Secondary Outcome: Pharmacodynamics of AZD9977 Assessed Per Total Sodium Excreted Cumulatively and During Each of the Urine Collection Intervals.
Description: Pharmacodynamics of AZD9977 by assessment of total sodium excreted cumulatively and during each of the urine collection intervals.
  Pharmacodynamics of AZD9977 after single dosing of AZD9977 with fludrocortisone and/or eplerenone.
Time Frame: From 0 to 24 hours after dosing
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mmol
Arm/Group | Treatment A | Treatment D | Treatment B | Treatment C
Number analyzed (Participants) | 23 | 23 | 23 | 23
mmol
  0 to 2 hours | 7 (3) | 8 (6) | 7 (3) | 7 (4)
  2 to 4 hours | 12 (6) | 17 (7) | 15 (5) | 15 (7)
  4 to 6 hours | 15 (8) | 31 (12) | 23 (8) | 23 (8)
  6 to 8 hours | 19 (10) | 46 (14) | 32 (10) | 34 (10)
  8 to 10 hours | 23 (12) | 63 (17) | 39 (12) | 47 (14)
  10 to 12 hours | 28 (14) | 74 (19) | 46 (13) | 55 (16)
  12 to 14 hours | 32 (17) | 82 (22) | 51 (14) | 62 (19)
  14 to 16 hours | 36 (18) | 87 (23) | 54 (15) | 67 (21)
  16 to 24 hours | 46 (23) | 103 (29) | 66 (19) | 79 (24)

24. Secondary Outcome: Pharmacodynamics of AZD9977 Assessed Per Fractional Potassium Excretion in Urine for Each Urine Collection Time Interval.
Description: Pharmacodynamics of AZD9977 assessed per fractional potassium excretion in urine for each urine collection time interval.
  Pharmacodynamics of AZD9977 after single dosing of AZD9977 with fludrocortisone and/or eplerenone
Time Frame: From 0 to 8 hours post dosing
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: % value
Arm/Group | Treatment A | Treatment D | Treatment B | Treatment C
Number analyzed (Participants) | 23 | 23 | 23 | 23
% value
  0 to 2 hours | 21.72 (6.49) | 22.19 (3.96) | 21.14 (5.74) | 21.66 (5.40)
  2 to 4 hours | 22.26 (4.22) | 20.30 (4.45) | 18.95 (2.78) | 21.15 (5.25)
  4 to 6 hours | 14.60 (3.19) | 12.49 (3.04) | 12.12 (3.03) | 12.48 (3.13)
  6 to 8 hours | 18.08 (4.64) | 13.35 (5.60) | 13.34 (4.56) | 13.48 (3.55)

25. Secondary Outcome: Pharmacodynamics of AZD9977 by Assessment of Total Potassium Excreted Cumulatively and During Each of the Urine Collection Intervals
Description: Pharmacodynamics of AZD9977 by assessment of total potassium excreted cumulatively and during each of the urine collection intervals.
  Pharmacodynamics of AZD9977 after single dosing of AZD9977 with fludrocortisone in comparison to AZD9977 placebo.
Time Frame: From 0 to 24 hours after dosing
Population: The PD analysis set will consist of all participants in the SAF with at least one evaluable sum of the logarithm of the sodium/potassium ratio from two hours up to eight hours post dose, and who have no major protocol deviations thought to impact on the analysis of the PD data.
Measure: Mean (Standard Deviation); unit: mmol
Arm/Group | Treatment A | Treatment D | Treatment B | Treatment C
Number analyzed (Participants) | 23 | 23 | 23 | 23
mmol
  0 to 2 hours | 13.6 (5.6) | 14.5 (3.1) | 14.0 (5.8) | 13.7 (4.2)
  2 to 4 hours | 29.0 (9.4) | 26.7 (5.7) | 27.1 (7.7) | 27.4 (7.6)
  4 to 6 hours | 38.3 (11.1) | 35.2 (6.8) | 35.5 (8.8) | 35.9 (9.2)
  6 to 8 hours | 49.9 (13.3) | 44.4 (8.7) | 44.6 (10.4) | 45.1 (10.7)
  8 to 10 hours | 61.4 (14.7) | 54.4 (10.2) | 53.8 (11.0) | 54.9 (11.0)
  10 to 12 hours | 71.1 (15.7) | 62.1 (12.2) | 63.3 (11.4) | 64.0 (12.4)
  12 to 14 hours | 80.7 (17.5) | 71.3 (15) | 72.5 (13.1) | 73.5 (12.6)
  14 to 16 hours | 87.7 (17.4) | 77.5 (15.1) | 79.2 (13.2) | 79.7 (12.9)
  16 to 24 hours | 101.8 (17.7) | 92.1 (13) | 94.4 (15.5) | 95.4 (12.0)

26. Secondary Outcome: Pharmacodynamics of AZD9977 Assessed Per Urine Production for Each Urine Collection Time Interval.
Description: Pharmacodynamics of AZD9977 assessed per urine production for each urine collection time interval.
  Pharmacodynamics of AZD9977 after single dosing of AZD9977 with fludrocortisone and/or eplerenone.
Time Frame: From 8 hours before dosing until 24 hours after dosing
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Treatment A | Treatment D | Treatment B | Treatment C
Number analyzed (Participants) | 23 | 23 | 23 | 23
mL
  -8 to -2 hours | 321.4 (208.3) | 309.3 (182.5) | 284.5 (186.4) | 294.9 (130.3)
  -2 to 0 hour | 303.5 (111.7) | 288.6 (99.3) | 274.3 (113.7) | 284.5 (90.2)
  0 to 2 hour | 307.4 (78.4) | 320.2 (102.6) | 305.0 (89.5) | 298.8 (68.9)
  2 to 4 hour | 272.2 (105.0) | 236.1 (80.1) | 245.6 (63.2) | 272.6 (85.8)
  4 to 6 hours | 178.8 (93.8) | 246.0 (115.7) | 229.9 (147.7) | 202.2 (99.5)
  6 to 8 hours | 216.6 (99.3) | 115.7 (121.6) | 273.6 (96.6) | 291.5 (135.5)
  8 to 10 hours | 266.0 (125.4) | 326.6 (111.7) | 246.6 (103.9) | 300.2 (121.1)
  10 to 12 hours | 337.1 (132.0) | 361.9 (149.0) | 309.0 (137.4) | 324.5 (143.6)
  12 to 14 hours | 280.2 (131.0) | 300.7 (141.8) | 306.0 (125.4) | 306.3 (152.2)
  14 to 16 hours | 357.3 (124.8) | 345.9 (129.0) | 326.5 (115.3) | 354.2 (138.6)
  16 to 24 hours | 296.0 (184.1) | 302.8 (181.1) | 292.2 (164.8) | 290.6 (90.2)

27. Secondary Outcome: Pharmacodynamics of AZD9977 by Assessment of Total Urine Volume Excreted Cumulatively and During Each of the Urine Collection Intervals
Description: Pharmacodynamics of AZD9977 by assessment of total urine volume excreted cumulatively and during each of the urine collection intervals.
  Pharmacodynamics of AZD9977 after single dosing of AZD9977 with fludrocortisone and/or eplerenone
Time Frame: From 8 hours before dosing until 24 hours after dosing
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Treatment A | Treatment D | Treatment B | Treatment C
Number analyzed (Participants) | 23 | 23 | 23 | 23
mL
  0 to 2 hour | 307.4 (78.4) | 320.2 (102.6) | 305.0 (89.5) | 298.8 (68.9)
  2 to 4 hour | 579.5 (127.2) | 556.3 (126.1) | 550.7 (109.2) | 571.4 (128.3)
  4 to 6 hours | 758.3 (186.3) | 802.2 (189.7) | 780.6 (204.6) | 773.6 (184.1)
  6 to 8 hours | 974.9 (235.6) | 1099.0 (199.1) | 1054.2 (201.4) | 1065.1 (261.1)
  8 to 10 hours | 1242.2 (288.9) | 1425.2 (235.6) | 1300.8 (192.6) | 1365.3 (261.1)
  10 to 12 hours | 1574.4 (329.0) | 1791.7 (283.6) | 1609.8 (264.2) | 1689.8 (300.9)
  12 to 14 hours | 1865.1 (378.9) | 2091.7 (354.6) | 1915.8 (264.2) | 1996.1 (330.7)
  14 to 16 hours | 2221.0 (340.7) | 2435.7 (304.4) | 2242.3 (233.3) | 2350.3 (316.6)
  16 to 24 hours | 2506.6 (388.6) | 2741.2 (293.9) | 2534.5 (236.3) | 2640.9 (347.5)

ADVERSE EVENTS:
Time Frame: SAEs will be collected from the signing of informed consent and AEs from randomization until post-study 5 to 7 days post-final study drug dose
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 2/23 | 3/23 | 2/23 | 4/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=23) | Treatment B (N=23) | Treatment C (N=23) | Treatment D (N=23)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distention (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Splinter (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a publication (e.g., in a scientific journal) based on the results of this study is envisaged, approval from AstraZeneca will be obtained and a draft manuscript will be submitted to AstraZeneca for scrutiny and comment. The choice of conduit will be mutually agreed on by the Principal Investigator and AstraZeneca.